CLINICAL TRIAL: NCT07005804
Title: Calcium Pyrophosphate Deposition (CPPD) Disease : Clinical and Paraclinical Profile, Gene Expression and Metabolomics of the Acute and Chronic Clinical Phenotype
Brief Title: Calcium Pyrophosphate Deposition (CPPD) Disease
Acronym: PYC-OMIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC-P00127
Record Dates: First submitted 2025-05-26; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Calcium Pyrophosphate Deposition Disease; Rheumatic Diseases
Keywords: Calcium pyrophosphate deposition disease; gene expression; acute clinical phenotype; chronic clinical phenotype; metabolic expression
MeSH Terms: conditions — Chondrocalcinosis; Rheumatic Diseases

STUDY DESIGN:
Intervention Model Description: The PYC-OMIC study is a prospective, single-centre, cross-sectional, comparative study of chronic versus acute forms of CPPD. It is an interventional study with minimal risks and constraints for chronic forms recruited prospectively. Acute forms are included retrospectively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a chronic CPPD (Experimental): Patients with diagnosis of chronic calcium pyrophosphate crystal arthritis (either acute recurrent or persistent arthritis), meeting the 2023 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) classification criteria, after evaluation by a rheumatologist from the rheumatology department.
  Interventions: Genetic: transcriptomic and metabolomic analysis

INTERVENTIONS:
Genetic: transcriptomic and metabolomic analysis — Venous blood samples for transcriptomic and metabolomic analysis will be taken in 3 x 4 mL ethylenediaminetetraacetic acid (EDTA) tubes and stored immediately at 4°C, before being cryopreserved at -80°C in 500 μL aliquots of plasma. In addition, for transcriptomic analysis, a sample will also be taken in a Paxgen RNA tube cryopreserved at -80°C.

SUMMARY:
The goal of this clinical trial is to describe the transcriptomic and metabolomic profile of patients with chronic Calcium Pyrophosphate Deposition (CPPD) compared to those with acute CPPD.

The hypotheses are as follows :

* It is hypothesised that there is a transcriptomic and metabolomic signature of CPPD which explains why therapeutic responses to different anti-inflammatory treatments differ from one phenotype to another one
* It is hypothesised that the acute and chronic clinical phenotypes of CPPD have different clinical, biological and imaging characteristics, as well as a differing predisposition toward crystalline deposition and inflammatory pathway activation.

The management of participants with chronic forms of the disease included in this research was modelled on the usual recommended management, including a biological workup, joint puncture, ultrasound and radiographic workup. Double-energy CT scans and transcriptomic and metabolomic analyses on plasma are not routine tests.

ELIGIBILITY:
Inclusion Criteria - Acute forms of CPPD: retrospective part of the study

* Cases included in the COLCHICORT cohort (NCT03128905), for whom this was the first acute episode of CPPD

Inclusion Criteria - Chronical forms of CPPD : prospective part of the study

* Patients affiliated to the French social security system
* Age ≥ 65 years
* Diagnosis of chronic CPPD (recurrent acute or persistent arthritis), meeting ACR/EULAR 2023,11 classification criteria after evaluation by a rheumatologist in the rheumatology department
* Progression of CPPD rheumatism for at least 3 months and still active CPPD rheumatism, defined by a visual analogue scale (VAS) of disease activity ≥ 40 and/or presentation of at least 1 crisis over the last 3 months
* Glomerular Filtration Rate (GFR) in Chronic Kidney Disease Epidemiology (CKD EPI Collaboration) ≥ 30ml/min/1.73m2
* Minimum time between the last intake of a crisis treatment and inclusion in the study, depending on their half-life, in order to not interfere with the results of the omics analyses: 2 weeks (Nonsteroidal Anti-Inflammatory Drugs Per Os (PO) or Intramuscular (IM) or Intravenous (IV); corticosteroids PO or IV; colchicine PO; anakinra Subcutaneous (SC), 1 month (methotrexate PO, tocilizumab SC), 3 months (canakinumab SC, tocilizumab IV)
* Signed written consent for study participation

Exclusion Criteria - Acute forms of CPPD:

* Missing data concerning transcriptomic and metabolomic analyses.
* Opposition

Exclusion Criteria - For chronic forms of CPPD:

* History of gout or presence of monosodium urate (MSU) crystals on joint fluid,
* Cognitive decline (confusion and neurodegenerative diseases)
* Inability to provide informed consent and disease VAS
* Patient under guardianship or curatorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Transcriptomic profile | 2 weeks
  -Quantitative transcriptomic profiling (expression of the genes involved) and qualitative profiling (analysis of the sequence of variants expressed)
Metabolomic profile | 2 weeks
  - Metabolomic profile: quantitative assessment of the metabolites involved in each phenotype, then qualitatively grouped by activated metabolic pathway

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte JAUFFRET, Principal Investigator — Rheumatology Department - Hôpital Saint-Vincent - GHICL
Locations (1):
- Hôpital Saint-Philibert (GHICL), Lomme, France

IPD SHARING:
Plan to Share IPD: No